CLINICAL TRIAL: NCT07225036
Title: PRIME-LRT: PRomoting IMmunotherapy Efficacy With Low-Dose Liver RT
Brief Title: Promoting Immunotherapy Efficacy With Low-Dose Liver RT
Acronym: PRIME-LRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Kharofa (Other)
Responsible Party: Sponsor-Investigator, Jordan Kharofa, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-RT-25-01
Record Dates: First submitted 2025-10-29; First posted 2025-11-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Low-Dose Liver Radiation (LD-LRT); Non Small Cell Lung Cancer; Melanoma; Liver Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Intervention Model Description: The trial will be conducted using Simon's optimal two-stage test in two separate cohorts. Cohort 1 will include patients with NSCLC with liver metastases. Cohort 2 will include patients with melanoma with liver metastases. The primary endpoint is 6-month PFS for each cohort compared separately to historical trials with an effect size goal of 25% improvement in 6-month PFS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LD-LRT (Experimental): Low-dose radiation to the liver the week prior to Cycles 1, 2 and 3 of systemic treatment.
  Interventions: Radiation: LD-LRT

INTERVENTIONS:
Radiation: LD-LRT — Low-dose radiation to the liver the week prior to Cycles 1, 2 and 3 of standard of care immunotherapy treatment.

SUMMARY:
The purpose of this study is to see if adding Low-Dose Liver Radiation (LD-LRT) improves progression free survival (PFS). This study is for patients with either melanoma or non-small cell lung cancer (NSCLC), with liver metastases, and receiving immunotherapy.

DETAILED DESCRIPTION:
Patients will continue standard of care immunotherapy (with or without standard chemotherapy). The research aspect of this study will be adding in the Low-Dose Liver Radiation (LD-LRT) before cycles 1, 2, 3 of treatment to see if this improves the treatment effects.

The trial will be conducted using Simon's optimal two-stage test in two separate cohorts. Cohort 1 will include patients with NSCLC with liver metastases. Cohort 2 will include patients with melanoma with liver metastases. The primary endpoint is 6-month PFS for each cohort compared separately to historical trials with an effect size goal of 25% improvement in 6-month PFS.

Cohort 1 NSCLC- The estimated 6-month PFS in NSCLC with liver metastasis was obtained from a metanalysis of 8 randomized trials evaluating the effect of liver metastases in patients treated with PD-1/PD-L1 inhibitors and chemotherapy (SOC) or chemotherapy alone[30]. Based on the pooled hazard ratios we estimate a 0.68 HR and PFS of 30% at 6 months with chemotherapy alone. Assuming underlining exponential distribution for survival time, we estimate the 6-month PFS is 44% in patients with liver metastases treated with PD-1/PD-L1 inhibitors and chemotherapy.

Simon's optimal two-stage design (Simon, 1989) will be used for conducting the trial. In cohort 1, the null hypothesis is that the true response rate (6-month PFS) is 0.44, and the alternative hypothesis is that the true response rate is 0.69. The trial is carried out in two stages. In stage I, a total number of 11 patients is accrued. If there are 5 or fewer responses among these 11 patients, cohort 1 will be stopped. Otherwise, an additional 15 patients will be accrued in stage II, resulting in a total number sample size of 26. If there are 16 or more responses among these 26 patients, we reject the null hypothesis and claim that the treatment is promising. The design controls the type I error rate at 0.049 and yields the power of 0.81. The probability of early termination is 66%.

Cohort 2 Melanoma with liver met (Expected 6-mo PFS= 30%, Desired 6-mo PFS=55%) The null hypothesis for 6-month PFS of 30%, based on historic clinical trials and series specifically evaluating PFS in patients with melanoma and liver metastases treated with standard of care immunotherapy[9-11, 14]. The alternative hypothesis is that the 6-month PFS is 55%. The trial is carried out in two stages. In stage I, a total number of 10 patients is accrued. If there are 3 or fewer responses among these 10 patients, the cohort will be closed. Otherwise, an additional 18 patients will be accrued in stage II for cohort 2, resulting in a total sample size of 28 patients. If there are 13 or more responses among these 28 patients, we reject the null hypothesis and claim that the treatment is promising. The design controls the type I error rate at 0.05 and yields the power of 0.8. The probability of early termination is 65%.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. ECOG performance status ≤2 (or Karnofsky ≥60%, see Appendix A).
3. Patients must have adequate organ and marrow function to receive standard of care immunotherapy and/or chemoimmunotherapy as per the treating medical oncologist.
4. Must be planning to, and able to, undergo active treatment with PD-L1 or PD-1 checkpoint immunotherapy given per standard care throughout the duration of the RT intervention per their treating physician.

   • Note: Patients may receive other SOC CTLA 4 inhibitors or other SOC chemotherapy/immunotherapy in combination with a SOC PD-L1 or PD-1 checkpoint inhibitor and remain eligible.
5. Biopsy proven Non-Small Cell Lung Cancer (NSCLC) or Melanoma.
6. Radiographic evidence of liver metastases.
7. Women of child-bearing potential and men must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
8. Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.
9. Patients must have insurance authorization to proceed with radiotherapy prior to initiation of radiation treatment on study

Exclusion Criteria:

1. Patients with prior immunotherapy use in the adjuvant setting for NSCLC or Melanoma are eligible unless the adjuvant immunotherapy was delivered within 6 months of enrollment.
2. Patients with NSCLC are ineligible for enrollment in cohort 1 if the presence of the following driver mutations are noted: EGFR, ALK, ROS1, RET.
3. Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous, in the opinion of the Investigator.
4. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen in the opinion of the Investigator.
5. Pregnant women are excluded from this study considering the use of ionizing radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) measured by 6-month PFS for each cohort compared separately to historical trials with an effect size goal of 25% improvement in 6-month PFS | 6 months
  The primary objective is to evaluate whether the addition of Low-Dose Liver Radiation (LD-LRT) improves progression free survival (PFS) in patients with melanoma and non-small cell lung cancer (NSCLC) with liver metastases receiving immunotherapy. The primary endpoint is 6-month PFS for each cohort compared separately to historical trials with an effect size goal of 25% improvement in 6-month PFS.

SECONDARY OUTCOMES:
Overall survival (OS) measured by time to death or last follow up | Enrollment to death or last follow-up (up to 2.5 years)
  The secondary objective is to evaluate whether the addition of Low-Dose Liver Radiation (LD-LRT) improves overall survival (OS) in patients with melanoma and non-small cell lung cancer (NSCLC) with liver metastases receiving immunotherapy. OS will be assessed as the time from enrollment to death or last follow-up.

OTHER OUTCOMES:
Immune profiling of patient peripheral blood mononuclear cells (PBMCs) | Baseline (Day -35), post-cycle 1 RT (Approx day 5), prior to cycle 2 RT (approx day 35), prior to cycle 3 RT (approx day 65), 3 months (approx day 90)
  1. To determine the immune profiling of patient peripheral blood mononuclear cells (PBMCs) for immunophenotype and activation status, and patient plasma for soluble immune/inflammatory mediators (i.e., cytokines) using flow cytometry-based and plasma based cytokine analysis.
TCR repertoire and clonal diversity in patients receiving LD-LRT and immunotherapy | Baseline (Day -35), post-cycle 1 RT (Approx day 5), prior to cycle 2 RT (approx day 35), prior to cycle 3 RT (approx day 65), 3 months (approx day 90)
  2. To evaluate T cell receptor (TCR) via TCR sequencing to characterize the TCR repertoire and clonal diversity in patients receiving LD-LRT and immunotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States